CLINICAL TRIAL: NCT02213991
Title: A Phase II Trial Investigating Acute Local Toxicities of Intraoperative Radiotherapy as a Boost Dose in Korean Breast Cancer Patients Undergoing Breast Conserving Surgery
Brief Title: Intraoperative Radiotherapy for Korean Patients With Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-IORT
Record Dates: First submitted 2014-08-05; First posted 2014-08-12 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Conservative Surgery; Intraoperative Radiotherapy; Local Toxicity; Whole breast radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Evaluate the safety of intraoperative radiotherapy using Intrabeam in Korean patients with early breast cancer.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative Radiotherapy (Experimental): Intervention:
  Intraoperative Radiotherapy
  * Operation day
  * Breast conservative surgery + Intraoperative radiotherapy 20 Gy
  Aftuer tumor lump is removed and negative tumor margins are achieved, applicator of Intrabeam® is located within tumor cavity. Purse string suture pulles up tissues and wraps up the applicator. IORT with 20Gy is followed. After IORT, applicator was out of the operative field, and usual wound closure will be done.
  * Postoperative period
  * ± Chemotherapy
  * WBRT (46 Gy) for 4~5 weeks
  * ± Endocrine therapy or target therapy
  Interventions: Device: Intraoperative radiotherapy using Intrabeam®

INTERVENTIONS:
Device: Intraoperative radiotherapy using Intrabeam® — Operation day
  1. Aftuer tumor lump is removed and negative tumor margins are achieved, applicator of Intrabeam® is located within tumor cavity.
  2. Purse string suture pulles up tissues and wraps up the applicator.
  3. Intraoperative radiotherapy using Intrabeam® (20Gy) is followed.
  4. After IORT, applicator was out of the operative field, and usual wound closure will be done.
     * Postoperative period
       * Chemotherapy WBRT (46 Gy) for 4~5 weeks
       * Endocrine therapy or target therapy

SUMMARY:
The purpose of this study is to evaluate acute local toxicity of IORT at the dose of 20 Gy for the replacement of boost-external beam radiotherapy in Korean women who are candidates for breast-conserving treatment.

DETAILED DESCRIPTION:
Local toxicity checklist

* Hematoma needing surgical evacuation
* Seroma needing more than three aspirations
* Skin breakdown or delayed wound healing
* Any complication needing surgical intervention
* Radiation Therapy Oncology Group (RTOG version 2.0) toxicity grade 3 or 4 for dermatitis, telangiectasia, pain in irradiated field, or other.
* Any complication of RTOG toxicity grade more than 2

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and newly diagnosed non-metastatic operable primary breast cancer
* Primary tumor <5cm, measured by ultrasonography - N0-3 (any N if resectable) and no evidence of distant metastasis (M) (isolated supraclavicular node involvement allowed)
* Age ≥18-years women with good performance status (ECOG 0-1)
* No breast operation is allowed except diagnostic biopsy
* Women with ductal carcinoma in situ diagnosed by preoperative biopsy are allowed

Exclusion Criteria:

* Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
* Patients who received prior chemotherapy or radiotherapy for breast cancer
* Patients who have history of cancer other than in situ uterine cervix cancer or non-melanoma skin cancer
* The depth of tumor from skin measured by ultrasonography is less than 1cm.
* Contraindications to breast conservative surgery

  * Multicentric breast cancer (tumors in more than one quadrant)
  * Diffuse malignant appearing microcalcification
  * Prior therapeutic radiation to the breast region
  * Small breast, which is not possible to achieve clear margins in relation to a cosmetically acceptable result
  * History of collagen vascular disease, such as active scleroderma and active lupus
* Postoperative exclusion

  * Patients who require re-excision due to positive resection margin
  * The depth of cavity from skin after lumpectomy is less than 0.5cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-08; Primary Completion 2017-10 (Actual); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Acute local toxicity in breast receiving IORT | Up to 6 months
  Acute local toxicities of ipsilateral breast occurred within 6 months after IORT
  Local toxicity checklist
  * Hematoma needing surgical evacuation
  * Seroma needing more than three aspirations
  * Skin breakdown or delayed wound healing
  * Any complication needing surgical intervention
  * Radiation Therapy Oncology Group (RTOG version 2.0) toxicity grade 3 or 4 for dermatitis, telangiectasia, pain in irradiated field, or other.
  * Any complication of RTOG toxicity grade more than 2
  Expected number of patients with acute local toxicites associated with IORT-booster treatement is 32.
  Considering a drop-out rate of 10%, the trial would need to enroll 215 patients in total.

SECONDARY OUTCOMES:
Delayed local toxicity | Up to 5 years
  Monitoring of local toxicity evaluated at 2 years and 5 years
Cosmesis | Up to 2 years
  Questionnaire on cosmetic outcome of operation site Qualified assessment based on BCCT ver 2.0
Local tumor recurrence in ipsillateral breast | Up to 5 years
  IBTR rate at 5 years
Dosimetray | At time of surgery
  -Dosimetry in tumor cavity and correlation with acute and late complication rates
  * Identification of anatomical indication
  * MRI volumetry (Breast-to-tumor ratio)
  * Skin depth measured at preoperative US

CONTACTS AND LOCATIONS:
Overall Officials: Joon Jeong, M.D. Ph.D., Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahn SG, Bae SJ, Lee HW, Yoon CI, Kim JW, Lee IJ, Jeong J. A phase II study investigating the acute toxicity of targeted intraoperative radiotherapy as tumor-bed boost plus whole breast irradiation after breast-conserving surgery in Korean patients. Breast Cancer Res Treat. 2019 Feb;174(1):157-163. doi: 10.1007/s10549-018-5038-x. Epub 2018 Nov 22. PMID 30467660